CLINICAL TRIAL: NCT03028324
Title: Investigating the Use of Transcranial Magnetic Stimulation (TMS) for Primary Progressive Apraxia of Speech (PPAOS)
Brief Title: Transcranial Magnetic Stimulation (TMS) for Primary Progressive Apraxia of Speech (PPAOS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting participants and lost personnel.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joyce Rios Gomes Osman, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20161125
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Apraxia Speech
MeSH Terms: conditions — Apraxias | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcranial Magnetic Stimulation (TMS) (Experimental): Non-invasive brain stimulation, high frequency repetitive TMS delivered in 10 sessions over a 2-week period.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Non-invasive brain stimulation, high frequency repetitive TMS delivered in 10 sessions over a 2-week period.

SUMMARY:
The purpose of this study is to assess the influence of transcranial magnetic stimulation (TMS) on speech performance in individuals with primary progressive apraxia of speech.

DETAILED DESCRIPTION:
Apraxia of speech (AOS) is a motor speech disorder affecting the programming of motor speech production. It is characterized by the impaired ability to coordinate the sequential, articulatory movements necessary to produce speech sound. It can result from insult to the brain, such as in stroke, or as the presenting sign/symptom of another neurodegenerative disease.

TMS is a neurostimulation technique which has been shown to modulate cortical excitability in a non-invasive manner, and has been associated with positive outcomes in a variety of neurological and psychological disorders.There is evidence to support the role of TMS in individuals with primary progressive aphasias. In addition, there is a a case report suggesting an improvement in speech following TMS in an individual with primary progressive AOS. This study is being undertaken to further examine the role of TMS in primary progressive AOS.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 and above who are able to consent
* Diagnosis of primary progressive apraxia of speech based on neurological evaluation

Exclusion Criteria:

* Any uncontrolled medical condition expected to limit life expectancy or interfere with participation in the trial (i.e. unstable cancer, severe depression or anxiety by DSM-IV criteria)
* Abnormal stress test, as determined by the treating physician (unless cardiology clearance provided)
* Active substance abuse or alcohol dependence
* Uncorrected vision or hearing deficits that would preclude administration of the cognitive measures
* Unwilling or unable to provide written informed consent
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or family history of treatment resistant epilepsy
* No medication is an absolute exclusion from TMS. Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following:

  * The subject's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other CNS active drugs.
  * The published TMS guidelines review medications to be considered with TMS
* Any metal in the brain, skull or elsewhere unless approved by the responsible MD
* Any medical devices (i.e. Cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator) unless otherwise approved by the responsible MD
* Substance abuse or dependence within the past six months
* Absence of corticospinal functional integrity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce R Gomes Osman, PT, PhD, Principal Investigator — Univeristy of Miami Miller School of Medicine
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Speech Performance
Description: Apraxia of Speech Rating Scale has a total range from 0-64, with lower scores indicating lower impairment and higher scores indicating higher impairment.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 4
score on a scale | -8.75 (8.06)

2. Secondary Outcome: Change in Motor Cortex Excitability
Description: Motor cortex excitability will be assessed with single-pulse TMS
Time Frame: Baseline, 4 weeks
Population: The change in motor excitability data is not available due to the fact that post intervention data was not collected.
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Transcranial Magnetic Stimulation (TMS)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT03028324/Prot_001.pdf